CLINICAL TRIAL: NCT00003124
Title: Phase II Trial of Maximal Androgen Deprivation Followed by Conformal External Beam Radiotherapy With Continued Androgen Deprivation for Clinically Localized Prostate Cancer
Brief Title: Hormone Therapy Plus Radiation Therapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065883; CPMC-IRB-7947; NCI-G97-1356
Record Dates: First submitted 1999-11-01; First posted 2003-04-18 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2002-12

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Flutamide; Leuprolide; Radiotherapy

INTERVENTIONS:
Drug: flutamide
Drug: leuprolide acetate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Androgens can stimulate the growth of prostate cancer cells. Hormone therapy using leuprolide and flutamide may fight prostate cancer by reducing the production of androgens. Combining radiation therapy with hormone therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of hormone therapy plus radiation therapy in treating patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the disease free survival of patients with localized adenocarcinoma of the prostate cancer.
* Evaluate the toxic effects of three dimensional conformal external beam radiotherapy and androgen deprivation in these patients.

OUTLINE: Patients are stratified according to PSA values and Gleason scores (class II versus class III/IV).

Patients receive intramuscular leuprolide acetate every 3 months, and oral flutamide tid.

Patients are evaluated on a monthly basis for response. Patients with unchanged or undetectable prostate specific antigen levels are considered to have reached maximal hormonal response and three dimensional conformal external beam radiotherapy is instituted. In addition, patients with disease progression are considered to have reached maximal response, and three dimensional conformal external beam radiotherapy is instituted. Radiotherapy must be administered within 6 months after initiation of leuprolide and flutamide therapy.

Hormonal therapy is administered until 9 months of treatment have elapsed.

Patients will be followed every 3 months for the first year, every 4 months for the second and third years, and every 6 months thereafter.

PROJECTED ACCRUAL: A total of 105 patients will be accrued from biologic class II over 3 years, and 58 patients from biologic class III-IV.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven localized adenocarcinoma of the prostate

  * Prostate specific antigen (PSA) greater than 4 or Gleason score at least 8 if PSA is no greater than 4
  * CT, MRI, or pelvic lymphadenectomy negative for metastases, if PSA is no greater than 50
  * Negative pelvic lymphadenectomy, if PSA is greater than 50
  * Bone scan negative for metastases or PSA no greater than 20

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance Status:

* Not specified

Life Expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm3
* Platelet count at least 70,000/mm3
* Hemoglobin at least 10 g/dL
* Patients on anticoagulant therapy must have a baseline PT test

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* ALT or AST less than 1.5 times ULN
* Alkaline phosphatase less than 1.5 times ULN

Renal:

* Creatinine less than 1.5 times ULN

Cardiovascular:

* No history of collagen vascular disease

Other:

* No acute infection requiring antibiotics
* No history of hypersensitivity to flutamide
* No history of hypersensitivity to leuprolide acetate

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 1997-05; Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald D. Ennis, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Heymann JJ, Benson MC, O'Toole KM, Malyszko B, Brody R, Vecchio D, Schiff PB, Mansukhani MM, Ennis RD. Phase II study of neoadjuvant androgen deprivation followed by external-beam radiotherapy with 9 months of androgen deprivation for intermediate- to high-risk localized prostate cancer. J Clin Oncol. 2007 Jan 1;25(1):77-84. doi: 10.1200/JCO.2005.05.0419. PMID 17194907